# Title of the study:

# Impact of biological factors on dental implant osseointegration

Study Number:

**MUOSU-202104.** 

Date: 6/9/2023

day / month / year



## **RESEARCH ETHICS: PATIENT INFORMATION FORM**

Study Number: MUOSU-202104

Title of Project: Impact of biological factors on dental implant osseointegration

## Principle investigator: Dr. Afya Sahib Diab

#### 1- What is the purpose of this study?

To develop the science of dental Implantology and find new ways to increase the success rates of dental implants

#### 2- Why have I been chosen?

You have missing teeth and you need dental implants to replace the missing teeth.

#### 3- Do I have to take part?

No, it's up to you

#### 4- What will happen to me if I take part?

Nothing will happen to you except you are going to help me carrying out my study research

#### 5- What are the possible disadvantages and risks of taking part?

There is no possible risk or disadvantage of taking part

#### 6- What are the possible benefits of taking part?

Taking part will facilitate my work during the research by collecting required number of cases needed which may provide beneficial treatment alternatives for you as well as others in the future

#### 7- Will my taking part in this study be kept confidential?

Sure, your information will be kept private

#### 8- What will happen to the results of the research study?

The results of the study research will be published in scientific magazines for the benefit of all

#### 9- Who is organizing & hosting the research?

Mustansiriyah University / College of dentistry

#### 10- What if I need more information about the way in which this study has been conducted?

You can ask your dentist about any information you need

Principal investigator: Dr. Afya Sahib Diab

Email: drafya\_diab@yahoo.com Phone No. +964(0)7816883387 Study Number: MUOSU-202104



| Patient identification number for this study: |
|---|
| Title of the Project: |
| Impact of biological factors on dental implant osseointegration |
| Principle investigator: Dr. Afya Sahib Diab |
| I. I confirm that I have read and understand the information sheet for the above study. I have had opportunity to consider the information, ask questions and have had these answered satisfactorily. |
| Consent form |
| <ul> <li>2. I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected.</li> <li>3. I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from regulatory authorities, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records.</li> <li>4. further samples may be taken during dental treatment as patients are being recruited at different time stage of treatment.</li> </ul> |
| I agree to take part in the above study |
| Name of the participant Date: day / month/ year Signature |
| Name of person taking consent Date: day/month/year Signature |